CLINICAL TRIAL: NCT01572649
Title: A Randomized, Double-blind, Placebo Controlled Trial to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Lixisenatide in Paediatric (10 - 17 Years Old) and Adult Patients With Type 2 Diabetes
Brief Title: Evaluation of the Blood Levels of the Drug (Lixisenatide), the Plasma Glucose Levels and Safety in Paediatric and Adult Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PKD11475; 2011-004584-67 (EudraCT Number); U1111-1124-3136 (Other: UTN)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 1 single administration (volume matched to the dose lixisenatide: 50 µL or 100µL) once a day subcutaneously
  Interventions: Drug: Placebo
- Dose 1 (Experimental): 1 single administration of 5 µg lixisenatide (50 µL) once a day subcutaneously
  Interventions: Drug: Lixisenatide (AVE0010)
- Dose 2 (Experimental): 1 single administration of 10 µg lixisenatide (100 µL) once a day subcutaneously
  Interventions: Drug: Lixisenatide (AVE0010)

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form:Solution for injection
  Route of administration: subcutaneous
  Arms: Dose 1; Dose 2
Drug: Placebo — Pharmaceutical form:Solution for injection
  Route of administration: subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

- To investigate the effects of two single subcutaneous lixisenatide doses (5 and 10 µg) as compared to placebo in reducing postprandial glucose (PPG) in type 2 diabetic paediatric population (10-17 years old) and adults as controls

Secondary Objectives:

- To evaluate in both paediatric and adult populations:

* the blood levels of lixisenatide (pharmacokinetic) parameters in plasma after single subcutaneous ascending doses
* the maximum post-prandial glucose excursion, and on the changes in insulin, C-peptide and glucagon plasma concentrations following a standardized breakfast
* safety and tolerability.

DETAILED DESCRIPTION:
The duration of the study for each patient is planned between 4 and 7 weeks including a screening period (25 to 30 days), 3 treatment periods 1-7 days apart, each period lasting only one day (Day 1) and an end-of-study visit between 1 to 7 days after the last dose administration.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients with type 2 diabetes mellitus, as defined by WHO (fasting plasma glucose ≥ 7 mmol/L (126mg/dL) or 2 hours postprandial plasma glucose ≥ 11.1 mmol/L (200 mg/dL)), diagnosed for at least 1 year (adults) and at least 3 months for paediatric population at the time of screening visit, with or without metformin (stable dose ± 10 % for at least 4 weeks prior to randomization)
* HbA1c ≥ 7% and ≤ 10% at screening
* Age eligibility for paediatric population: ≥ 10 years and <18 years with at least 3 patients below 15 years and no more than 3 patients aged between 16 and 18 years; Age eligibility for adults: ≥ 18 and ≤ 65 years
* For paediatric population:body weight >50kg, BMI >85th percentile for age and gender and BMI ≤ 50 kg/m²
* For adults: BMI > 25 kg/m2 and ≤ 37 kg/m2

Exclusion criteria:

* If female, pregnancy (defined as positive serum pregnancy test), breast-feeding
* Diabetes other than type 2 diabetes
* Positive test for insulinoma associated protein (IA2) and glutamic acid decarboxylase (GAD) autoantibodies
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin (e.g., alpha glucosidase inhibitor, exenatide, DPP-IV inhibitors, insulin etc.) within 3 months prior to the time of screening
* Allergic reaction to any GLP-1 agonist in the past (e.g. exenatide, liraglutide) or to metacresol
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease
* Personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (e.g., multiple endocrine neoplasia syndromes)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
GLU-AUC 0:30-4:30h: area under the plasma glucose concentration time profile from time of the standardized breakfast start (30 min after IMP injection and pre-meal plasma glucose) until 4 hours later subtracting the pre-meal value | D1 at each period up to 4h30 after study drug injection (8 timepoints)

SECONDARY OUTCOMES:
Pharmacokinetics: lixisenatide plasma concentration | 0 (predose), 30 min, 1h, 1h30, 2h30, 3h30, 4h30 and 6h30 post-dose at D1 of each study period (8 timepoints)
Pharmacokinetic parameter (Cmax) | calculated over the period of timepoints at D1 of each study period
Pharmacokinetic parameter (Tmax) | calculated over the period of timepoints at D1 of each study period
Pharmacokinetic parameter (AUC last) | estimated over the period of timepoints at D1 of each study period
Pharmacokinetic parameter (AUC) | extrapolated based on the period of timepoints at D1 of each study period
Area under the concentration time profile from time of standardized breakfast start (30 min after IMP injection) until 4 hours later for insulin, C-peptide and glucagon | D1 at each period up to 4h30 after study drug injection (7 timepoints)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (3):
  - Investigational Site Number 840005, Chula Vista, California
  - Investigational Site Number 840001, Overland Park, Kansas
  - Investigational Site Number 840003, Louisville, Kentucky
- Investigational Site Number 484001, Puebla City, Mexico
- Investigational Site Number 710002, Cape Town, South Africa
- Investigational Site Number 826001, Leeds, United Kingdom